CLINICAL TRIAL: NCT02479607
Title: PhONEME - ParticipatOn Ehealth MobilE. Effects of an Interactive ICT-platform for Assessment and Management of Symptoms in Patients Treated for Breast Cancer.
Brief Title: Effects of an ICT-platform for Assessment and Management of Patient-reported Symptoms During Treatment for Breast Cancer
Acronym: PhONEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Ann Langius-Eklöf, RN, PhD, Professor, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PhONEME Breast
Record Dates: First submitted 2015-06-12; First posted 2015-06-24 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Cytostatic Agents; Nursing; Health Literacy; Quality of Life; Oncology Nursing; Self Care; Symptom Management; Participatory Care; Person-centered Care; Information and Communication Technology; Patient-reported symptoms; Mobile device
MeSH Terms: conditions — Breast Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Use of an application for a smartphone or tablet for daily reporting symptoms and access to self-care advice and health care professionals in real time in combination with standard care according to the clinic´s routines
  Interventions: Device: Smartphone or tablet
- Control group (No Intervention): Standard care according to the clinic's routines.

INTERVENTIONS:
Device: Smartphone or tablet
  Other Names: Intervention
  Arms: Intervention group

SUMMARY:
The purpose of this study is to evaluate the effects of an interactive Information and Communication Technologies (ICT) -platform for use in a smartphone or tablet in patients treated with neoadjuvant chemotherapy for breast cancer. The hypothesis is that clinical management will be improved and costs reduced and safe and participatory care promoted, when patients report symptoms in an application which provides self-care advice and instant access to professionals.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of breast cancer
* Patients who will receive neoadjuvant chemotherapy
* Literacy in the Swedish language

Exclusion Criteria:

* Patients who need an interpreter at the doctor's visit
* Patients who have a known severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Questionnaire Scale for Functional Health Literacy (S-FHL-Swedish version) | Up to 3 months after completion of neoadjuvant chemotherapy treatment
  To evaluate self-reported data in terms of understanding health
Questionnaire Scale for Communicative and Critical Health Literacy (S-C & C HL - Swedish version) | Up to 3 months after completion of neoadjuvant chemotherapy treatment
  To evaluate self-reported data in terms of communicating health
Questionnaire Individualized Care Scale (ICS) | Up to 3 months after completion of neoadjuvant chemotherapy treatment
  To evaluate self-reported data in terms of individualized care
Questionnaire Sense of Coherence Scale (KASAM) | Up to 3 months after completion of neoadjuvant chemotherapy treatment
  To evaluate self-reported data in terms of Sense of Coherence
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) | Up to 3 months after completion of neoadjuvant chemotherapy treatment
  To evaluate self-reported data in terms of health related quality of life
Questionnaire Memorial Symptom Assessment Scale (MSAS) | Up to 3 months after completion of neoadjuvant chemotherapy treatment
  To evaluate self-reported data in terms of symptom prevalence, characteristics and distress

SECONDARY OUTCOMES:
Health care costs | Up to 3 months after completion of neoadjuvant chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ann Langius-Eklöf, RN, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Crafoord MT, Ekstrand J, Sundberg K, Nilsson MI, Fjell M, Langius-Eklof A. Mobile Electronic Patient-Reported Outcomes and Interactive Support During Breast and Prostate Cancer Treatment: Health Economic Evaluation From Two Randomized Controlled Trials. JMIR Cancer. 2025 Mar 11;11:e53539. doi: 10.2196/53539. PMID 40067346
- [Derived] Langius-Eklof A, Crafoord MT, Christiansen M, Fjell M, Sundberg K. Effects of an interactive mHealth innovation for early detection of patient-reported symptom distress with focus on participatory care: protocol for a study based on prospective, randomised, controlled trials in patients with prostate and breast cancer. BMC Cancer. 2017 Jul 4;17(1):466. doi: 10.1186/s12885-017-3450-y. PMID 28676102